CLINICAL TRIAL: NCT03479411
Title: Phase 1, 3-Part, Open-Label Study to Assess Safety, Tolerability and PK of Single and Multiple Doses of PUR1900 in Healthy Subjects and Crossover Study of Single Doses of PUR1900 and Sporanox in Adult Subjects With Mild to Moderate Asthma
Brief Title: Safety, Tolerability and Pharmacokinetics of PUR1900 (Itraconazole Powder) in Healthy Volunteers and Adults With Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pulmatrix Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 601-0013
Record Dates: First submitted 2018-02-05; First posted 2018-03-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Itraconazole

STUDY DESIGN:
Intervention Model Description: The study has 3 parts: 1) Single Ascending Dose Escalation and 2) Multiple Ascending Dose Escalation to be conducted in Normal Healthy Volunteers and 3) A two-period crossover study of single doses of PUR1900 and Sporanox in Adults with Asthma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1 single ascending dose (Experimental): Intervention: drug Itraconzaole powder: single dose of 5mg, 10mg or 25 mg Other name: PUR1900
  Interventions: Drug: Itraconazole Powder
- Part 2 multiple ascending dose (Experimental): Intervention: drug Itraconzaole powder: 10 mg or 20 mg daily for 14 days Other name: PUR1900
  Interventions: Drug: Itraconazole Powder
- Part 3 2-period crossover single dose (Active Comparator): Intervention: drug Itraconzaole powder: 20 mg single dose and Itraconzaole oral solution 200 mg single dose Other names: PUR1900, Sporanox
  Interventions: Drug: Itraconazole Powder; Drug: Itraconazole 200 mg

INTERVENTIONS:
Drug: Itraconazole Powder — Itraconazole administered as a dry powder for inhalation (PUR1900)
  Other Names: PUR1900
Drug: Itraconazole 200 mg — Sporanox® Oral Solution
  Other Names: Sporanox®
  Arms: Part 3 2-period crossover single dose

SUMMARY:
Phase 1, 3-part study to assess safety, tolerability and PK of single and multiple doses of itraconazole administered as a dry powder for inhalation (PUR1900) in healthy subjects (parts 1 and 2) and a 2-period crossover study of single doses of itraconazole administered as a dry powder for inhalation (PUR1900) and an oral solution (Sporanox) in adults with mild to moderate, stable asthma (part 3)

DETAILED DESCRIPTION:
Phase 1, multi-center, 3-part, open-label study in healthy adults (Parts 1 and 2) and adults with mild to moderate, stable asthma (Part 3).

Safety, tolerability and PK will be assessed following either single ascending (SAD) or multiple ascending (MAD) dosing of itraconazole administered as a dry powder for inhalation (PUR1900; Part 1 and Part 2, respectively). Part 1 will comprise 3 separate cohorts planned to receive single doses of 5, 10 and 25 mg itraconzaole, respectively. The study will have an interleaved design; Part 2 will comprise 2 separate cohorts planned to receive daily doses of itraconazole 10 and 20 mg per day for 14 days, respectively. Part 2, Cohort 1 will commence after a review of safety data from Part 1 Cohort 2 suggests it is safe to do so.

Part 3 is a 2-period, randomised, crossover study in adult subjects with mild to moderate stable asthma to assess the safety, tolerability and PK of single doses of itraconazole administered as a dry powder for inhalation (PUR1900) and administered as an oral solution (Sporanox® Oral Solution).

ELIGIBILITY:
Inclusion Criteria:

Part 1 (SAD) and Part 2 (MAD):

1. Healthy males or non-pregnant, non-lactating healthy females.
2. Age 18 to 60 years
3. Screening forced expiratory volume in 1 sec (FEV1) ≥80% of the predicted value
4. Screening FEV1/forced vital capacity (FVC) >0.70.
5. Able to demonstrate the correct inhalation technique for use of delivery device during the study.

Part 3 (Asthmatic Subjects):

1. Males or non-pregnant, non-lactating females with a physician-confirmed diagnosis of asthma for at least 3 months. Asthma must be assessed by investigator as being stable for at least 4 weeks prior to screening.
2. Age 18 to 60 years
3. Subject is being treated with either inhaled corticosteroids (ICS) or inhaled corticosteroids plus long-acting beta-agonists (ICS/LABA). Only GINA STEP 2 and 3 patients will be enrolled.
4. Pre-bronchodilator, clinic measured, FEV1 ≥70% of predicted normal at screening
5. Able to perform the required spirometric testing.
6. Able to produce a sputum sample of a quality required for drug concentration assessments (a single repeat is permitted).

Exclusion Criteria:

1. Subjects who have received any IMP in a clinical research study within the previous 3 months prior to dosing on this study
2. Subjects who have previously received IMP in this study. Subjects who have participated in Part 1 are not permitted to participate in Part 2 or Part 3.
3. History of any drug or alcohol abuse in the past 2 years prior to screening.
4. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
5. Females of childbearing potential who are pregnant or lactating, or who plan to become pregnant during the study (all female subjects must have a negative pregnancy test at screening). A woman is considered of childbearing potential unless she is permanently sterile (hysterectomy, bilateral salpingectomy, bilateral oophorectomy, bilateral tubal occlusion/ligation) or is postmenopausal (had no menses for 12 months without an alternative medical cause (will be re-assessed at admission/pre-dose).
6. Positive drugs of abuse test result at screening or admission
7. Subjects with congestive heart failure or a history of congestive heart failure
8. History of severe cough or bronchospasm upon inhalation of any dry powder inhalation product
9. Subjects who are taking or have taken any herbal remedies or CYP3A4 inducers in the 28 days prior to the first IMP administration
10. Upper respiratory tract infection (excluding otitis media), fever, acute or chronic cough within 14 days of the first IMP administration, or lower respiratory tract infection within the last 3 months prior to IMP administration
11. Recent (last 4 weeks prior to IMP administration) clinically significant bacterial, viral or fungal infection that required systemic (oral or intravenous) antibiotics, antivirals or antifungals; topical treatments, other than antifungals, are allowed.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related Adverse Events as assessed by CTCAE v4.0 | Part 1: Baseline through Day 14, Part 2 and 3: Baseline through Day 28
  Safety and tolerability will be assessed by evaluating the number of participants with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Area under the serum concentration vs time curve from time 0 to infinity (AUC0-inf) of single dose of itraconazole | Part 1: Baseline through Day 14, Part 2 and 3: Baseline through Day 28
  The area under the serum concentration vs time curve from time 0 to infinity (AUC0-inf)
Time of the maximum measured serum concentration (Tmax) of single dose of itraconazole | Part 1: Baseline through Day 14, Part 2 and 3: Baseline through Day 28
  Time of the maximum measured serum concentration (Tmax)
Area under the serum concentration vs time curve within the dosing interval (AUCtau) of single dose of itraconazole | Part 1: Baseline through Day 14, Part 2 and 3: Baseline through Day 28
  The area under the serum concentration vs time curve within the dosing interval (AUCtau)
Apparent first-order terminal elimination half-life (t1/2 ) of single dose of itraconazole | Part 1: Baseline through Day 14, Part 2 and 3: Baseline through Day 28
  Apparent first-order terminal elimination half-life (t1/2 )
Apparent first-order terminal elimination rate constant calculated from a semi-log plot of the serum concentration vs time curve (Kel) of single dose of itraconazole | Part 1: Baseline through Day 14, Part 2 and 3: Baseline through Day 28
  Apparent first-order terminal elimination rate constant calculated from a semi-log plot of
Apparent clearance (CL/F) of single dose of itraconazole | Part 1: Baseline through Day 14, Part 2 and 3: Baseline through Day 28
  Apparent clearance (CL/F)
Apparent volume of distribution (Vz/F) of single dose of itraconazole | Part 1: Baseline through Day 14, Part 2 and 3: Baseline through Day 28
  Apparent volume of distribution (Vz/F)

OTHER OUTCOMES:
Maximum Concentration [Cmax] of itraconazole and hydroxyitraconazole in sputum | Part 3: baseline through 28 days
  Exploratory objective: To characterize the concentrations of itraconazole in induced sputum after single doses of inhaled PUR1900 and oral Sporanox® solution in subjects with mild to moderate stable asthma
Area under the Curve [AUC] of itraconazole and hydroxyitraconazole in sputum | Part 3: baseline through 28 days
  Exploratory objective: To characterize the concentrations of itraconazole in induced sputum after single doses of inhaled PUR1900 and oral Sporanox® solution in subjects with mild to moderate stable asthma

CONTACTS AND LOCATIONS:
Overall Officials: James Roach, MD, Study Director — Pulmatrix Inc.
Locations (2):
- United Kingdom (2):
  - Medicines Evaluation Unit, Manchester
  - Quotient Sciences, Nottingham

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bergagnini-Kolev M, Kane K, Templeton IE, Curran AK. Evaluation of the Potential for Drug-Drug Interactions with Inhaled Itraconazole Using Physiologically Based Pharmacokinetic Modelling, Based on Phase 1 Clinical Data. AAPS J. 2023 Jun 21;25(4):62. doi: 10.1208/s12248-023-00828-z. PMID 37344751